CLINICAL TRIAL: NCT07137156
Title: Metagenomic Analysis of the Oral Microbiome in Patients With Oral Lichen Planus: A Pilot Study
Brief Title: Metagenomic Analysis of the Oral Microbiome in Patients With Oral Lichen Planus: A Pilot Study in the Turkish Population
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, AYŞE GÜL ÖNER TALMAÇ, Assistant Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: AysegulOralLichen
Record Dates: First submitted 2025-08-06; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Oral Lichen Planus
Keywords: oral microbiome; NGS; oral lichen planus; metagenomic analysis
MeSH Terms: conditions — Lichen Planus, Oral | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- oral lichen planus: buccal smear
  Interventions: Diagnostic Test: cytobrush; Device: next-generation sequencing
- oral lichen planus healty: buccal smear
  Interventions: Device: next-generation sequencing
- control: buccal smear
  Interventions: Device: next-generation sequencing

INTERVENTIONS:
Diagnostic Test: cytobrush — buccal smear
  Groups: oral lichen planus
Device: next-generation sequencing — next-generation sequencing

SUMMARY:
Lichen planus is a common chronic mucocutaneous inflammatory disease that affects the skin, nails, eyes, urogenital system, and oral mucosa. Oral lichen planus (OLP) specifically occurs in the oral cavity. As a variant of lichen planus, OLP is believed to affect the oral mucosa through T-cell-mediated chronic inflammation, and some researchers suggest that Th2-mediated inflammation may also contribute to its pathogenesis. The absence of metagenomic analyses targeting oral microbiome profiling in OLP patients in Türkiye highlights the need for studies in this field. This pilot study, conducted for the first time in Türkiye, examined microbial diversity and dominant bacterial families in the lesional and non-lesional oral sites of Turkish individuals with OLP, compared with healthy individuals. The findings are expected to contribute to identifying potential microbial targets that may play a role in OLP pathogenesis and to shaping future treatment strategies.

DETAILED DESCRIPTION:
Lichen planus is a chronic dermatological disease. It is characterized by papules that are localized in areas exposed to mechanical irritation, mostly in areas of friction from clothing, on the inner and back parts of the legs, on the inner parts of the forearms, and on the wrists. It usually manifests itself as itching on the skin. Lichen planus can be observed in 40% of cases in both the skin and oral mucosa, 35% in the skin, and 25% only in the oral mucosa. In oral lichen planus (OLP), unlike in the skin, itching does not occur. Lesions in the oral mucosa appear as white, non-exfoliating, keratinized epithelial changes consisting of fine lines resembling a net or leaf veins, surrounded by erythema. Lesions are generally asymptomatic, but different types may present with symptoms such as pain or burning.

Andreassen (21) classified the clinical types of OLP as follows:

1. Reticular: Characterized by small gray-white papules that do not separate from the mucosa when wiped. They are typically located on the cheek mucosa and are symmetrical. These papules may have a thin erythematous border, and these formations often resemble a net or leaf veins (Wickham's lines).
2. Papular: Fine, linear extensions are seen around white hyperkeratotic formations that are 0.5-1 mm in diameter and raised above the surface.
3. Hypertrophic: These are dense white formations that are raised above the surface, particularly seen in smokers. Clinically, this type of OLP is difficult to distinguish from leukoplakia. Wickham's lines around the lesion may aid in establishing a preliminary diagnosis of lichen planus.
4. Atrophic: In this type, erythema is prominent and there is thinning of the epithelium. Those localized in the gingiva may transform into pemphigoid gingivitis. It may occur in conjunction with erosive and bullous OLP. This type may show a possibility of malignant formation. e. Erosive: This is the most common clinical type of OLP, characterized by erosions covered with dense fibrin and shallow ulcers. Erosions cause a burning sensation in OLP patients. This complaint may increase with mechanical, chemical, and thermal irritation associated with food intake.

Despite significant efforts over the past two decades to determine the etiology of OLP, the exact mechanism remains unclear. Previous studies have shown that T cells are involved in the pathogenesis of the disease, but their specific roles in this process remain unclear. Generally, an exogenous antigen, autoantigen, or superantigen triggers an inflammatory response leading to apoptosis of basal epithelial keratinocytes in the oral epithelium, resulting in chronic inflammation. A more plausible theory suggests that multiple antigens, combined with various environmental factors, trigger an inflammatory process. Therefore, the etiology is expected to be multifactorial, as in many other diseases, rather than a single causal factor, which is the approach most researchers use to study OLP.

Studies specific to OLP have shown that rigorous oral hygiene and plaque control can improve gingival lichen planus lesions, suggesting that the oral microbiome may play a role in the onset or exacerbation of OLP. The role of the oral microbiome has also been examined in other inflammatory oral mucosal disorders, such as recurrent aphthous stomatitis and geographic tongue, as well as in other autoimmune diseases, including Sjögren's syndrome, rheumatoid arthritis, and systemic lupus erythematosus. Additionally, recent studies on burning mouth syndrome have also shown that the oral microbiome is effective. Although the exact role of the oral microbiome in the pathogenesis of these conditions remains unclear, it can be suggested that it may also play a role in OLP.

Studies on the relationship between oral bacteria and OLP are available. He et al., in their study evaluating the bacterial composition of the buccal mucosa in patients with oral lichen planus, collected buccal swab samples from 43 patients with oral lichen planus (21 erosive and 22 non-erosive) and 21 healthy mucosal volunteers, and found that 94.26% of the total bacteria were classified into 15 genera present in large quantities. In all cases, Streptococcus, Prevotella, Haemophilus, Neisseria, Fusobacterium, Leptotrichia, Veillonella, and Actinomyces species were detected. In the study, Streptococcus was more prevalent in the healthy control group (p <0.01), while Fusobacterium (p < 0.01), Leptotrichia (P < 0.001), and Lautropia (P < 0.001) were more prevalent in the OLP group.

Compared to healthy control subjects, studies have shown that there is dysbiosis in the mucosal bacterial composition and salivary microbiota in OLP patients, and that there is a difference between affected and unaffected areas in the same patient. The literature also reports that certain species damage the epithelial barrier, invade the lamina propria, and internalize epithelial cells or T cells, leading to the production of specific T-cell chemokines.

The aim of this study was to determine the metagenomic profile analysis of relevant oral pathogens in patients with oral lichen planus.

ELIGIBILITY:
Inclusion Criteria:

* • Individuals who agree to participate in the study,

  * Aged between 18 and 75,
  * Individuals with OLP that has clinical and histopathological characteristics according to the World Health Organization FOR HEALTHY INDIVIDUALS; CRITERIA FOR PARTICIPATION IN THE STUDY
  * Individuals who agree to participate in the study,
  * Aged between 18 and 75,
  * Healthy individuals with no systemic disorders

Exclusion Criteria:

* • Individuals with oral mucosal diseases other than OLP,

  * Individuals with systemic disorders (autoimmune diseases, hematological diseases, diabetes mellitus, hypertension, infectious diseases, allergic conditions),
  * Use of systemic or topical medication for OLP within the last six months, FOR HEALTHY INDIVIDUALS;

CRITERIA FOR EXCLUSION FROM THE STUDY

• Individuals with OLP and other autoimmune-related oral mucosal diseases,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group consisted of 7 patients who applied to the Department of Oral and Maxillofacial Radiology Clinic of the Faculty of Dentistry at Marmara University and were clinically and histopathologically diagnosed with "OLP" (mucosa with OLP lesions and healthy mucosal tissue from the same patient). while 6 individuals who presented to our clinic for any complaint, were healthy, and agreed to participate in the study, and who did not have any autoimmune-related complaints, will form the control group.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
patient selection and sample collection | 1 month
  A 50 mg tissue sample will be collected from the patients using a cytobrush and transferred to 2.0 ml centrifuge tubes. The tubes will be stored at -80°C for DNA isolation.
DNA isolation | 2 week
  DNA extraction will be performed as a service purchase using the QIAmp DNA Mini Kit (Qiagen) with the QIACube Lt automated isolation device according to the manufacturer's protocol. A 50 mg tissue scraping sample will be homogenized in 200 μL of 0.9% NaCl before adding proteinase K and lysis buffer, following the Purelink protocol. Isolated DNA will be measured using a QIAxpert Nanospectrophotometer (A260) at absorbance. If DNA amounts exceed 30 ng/μl, samples will be sent for microbiota analysis.
Microbiota analysis | 2 month
  Sequencing was performed using the Illumina iSeq100 platform. In the bioinformatic analysis of raw data, fastq files were classified into OTU categories using the Kraken metagenomic system.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayşe Gül Öner Talmaç, Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT07137156/Prot_SAP_ICF_000.pdf